CLINICAL TRIAL: NCT02060591
Title: Comparison of Two Periarticular Injection Medications for Adjunctive Pain Management Following Total Knee Arthroplasty (TKA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 14PAR01
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Bupivacaine

ARMS (2):
- Exparel (Active Comparator)
  Interventions: Drug: Exparel
- Marcaine (Active Comparator)
  Interventions: Drug: Marcaine

INTERVENTIONS:
Drug: Exparel
  Arms: Exparel
Drug: Marcaine
  Arms: Marcaine

SUMMARY:
The Investigators aim to study the efficacy of Exparel as compared to Marcaine, taking into account pain control, narcotic consumption, narcotic-related side effects, outcomes measures, and patient satisfaction. Moreover, the Investigators plan to perform cost-benefit analysis to evaluate whether use of Exparel decreases analgesic consumption, duration of hospital stay and the need for physical therapy postoperatively, therefore, offsetting its higher price in comparison with Marcaine.

ELIGIBILITY:
Inclusion Criteria:

All patients at least 18 years old who have primary unilateral TKA for osteoarthritis performed at Thomas Jefferson University Hospital.

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) score of 4 or higher
* Hepatic disease (contraindication for acetaminophen)
* Renal disease (contraindication for NSAIDs)
* Any contraindication for oxycodone, ketorolac, epinephrine, pregabalin, gabapentin, hydromorphone, Tramadol, morphine or other narcotics that are considered as part of routine postoperative pain control protocol
* Fibromyalgia
* Any contraindication for intrathecal opioid injection
* History of substance abuse during the last 2 years
* History of allergy to amide compounds
* Current consumption of monoaminoxidase (MAO) inhibitors and tricyclic antidepressant (TCA) medications
* Allergy to metabisulfite compounds
* Chronic use of opioid medications in the month prior to surgery (leads to opioid tolerance and/or opioid-induced hyperalgesia)
* Body weight<50 Kg, BMI>40 Kg/m2
* History of hypotension
* Patients with any surgery related complication in the first 4-6 weeks following TKA, such as infection or mechanical failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
2. Measure pain intensity score (pre and post-operatively) by visual analogue scale (VAS) method | Within first 30 days post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Alijanipour P, Tan TL, Matthews CN, Viola JR, Purtill JJ, Rothman RH, Parvizi J, Austin MS. Periarticular Injection of Liposomal Bupivacaine Offers No Benefit Over Standard Bupivacaine in Total Knee Arthroplasty: A Prospective, Randomized, Controlled Trial. J Arthroplasty. 2017 Feb;32(2):628-634. doi: 10.1016/j.arth.2016.07.023. Epub 2016 Aug 9. PMID 27667533